CLINICAL TRIAL: NCT04231591
Title: NT-proBNP Levels in the Prediction of Intrapartum and Postpartum Events in Adult Congenital Heart Disease Patients
Acronym: NT-proBNP
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Carl H. Rose, Principal Investigator, Mayo Clinic
Other Study IDs: 19-005429
Record Dates: First submitted 2019-11-12; First posted 2020-01-18 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Congenital Heart Disease; Pregnancy Complications
MeSH Terms: conditions — Heart Defects, Congenital; Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACDH Pregnancy - Study group: Pregnant women with known adult congenital heart disease.
  Interventions: Diagnostic Test: NT-proBNP
- Uncomplicated pregnancy - Control group: Healthy women with an uncomplicated pregnancy
  Interventions: Diagnostic Test: NT-proBNP

INTERVENTIONS:
Diagnostic Test: NT-proBNP — Collect serum NT-proBNP levels in singleton ACHD patients and a comparative normotensive control group at time of admission for delivery to characterize negative predictive values for intrapartum and postpartum cardiac events.

SUMMARY:
The purpose of this study is to determine if NT-BNP levels obtained at time of admission for delivery are predictive of intrapartum or postpartum complications in patients with adult congenital heart disease.

DETAILED DESCRIPTION:
Amino-terminal pro-B-type natiuretic peptide (NT-proBNP) is a prohormone released from cardiac ventricular myocytes in direct response to cardiac workload. Secreted in the biologically inactive form, NT-proBNP is cleaved in the circulation into BNP, which subsequently exerts both vasodilatory and diuretic effects. The principal clinical utility of serum NT-proBNP measurement has been as an adjunctive marker in the diagnosis of subclinical heart failure, with higher levels typically reflective of increasing cardiac dysfunction.

The proposed prospective cohort study intends to collect serum NT-proBNP levels in singleton ACHD patients and a comparative normotensive control group at time of admission for delivery to characterize negative predictive values for intrapartum and postpartum cardiac events. Both pregnant patients with previously-diagnosed ACHD and those diagnosed and delivering during the study interval will be candidates for participation, and a gestational age threshold of 37 weeks will be utilized for the control group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant adult women ages 18 - 50
* Pregnancy with congenital heart disease (study group) or without congenital heart disease (control group)

Exclusion Criteria:

* Non-pregnant patients
* Non-English-speaking patients
* Maternal age <18 years or >50 years
* Patients with hypertensive complications of pregnancy
* Maternal peripartum cardiomyopathy
* Multiple gestation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females
Study Population: This study intends to collect serum NT-proBNP levels in singleton ACHD patients and a comparative normotensive control group at time of admission for delivery to characterize negative predictive values for intrapartum and postpartum cardiac events. Both pregnant patients with previously-diagnosed ACHD and those diagnosed and delivering during the study interval will be candidates for participation. A gestational age threshold of 37 weeks will be utilized for the control group.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Intrapartum cardiac complications | Inpatient admission for subsequent 48 hours
  Incidence of heart failure, incidence of arrhythmia, incidence of cardiac arrest
Postpartum cardiac complications | Initial 96 hours following delivery of infant(s)
  Incidence of heart failure, incidence of arrhythmia, incidence of cardiac arrest

SECONDARY OUTCOMES:
Intrapartum obstetrical complications | Inpatient admission for subsequent 48 hours
  Incidence of preeclampsia or gestational hypertension, incidence of placental abruption, cesarean section rate
Postpartum obstetrical complications | Initial 96 hours following delivery of infant(s)
  Incidence of postpartum hemorrhage, incidence of venous thromboembolism

CONTACTS AND LOCATIONS:
Overall Officials: Carl H. Rose, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20473511